CLINICAL TRIAL: NCT06335355
Title: A Phase II/III, Randomized, Open-label, Parallel-controlled, Multicenter Study of Adebrelimab (SHR-1316) in Combination With SHR-8068 and Platinum-based Doublet Chemotherapy as First-line Treatment in Advanced or Metastatic NSCLC Patients With STK11/KEAP1/KRAS Mutations
Brief Title: A Phase II/III Study of Adebrelimab in Combination With SHR-8068 and Chemotherapy in Advanced or Metastatic NSCLC Patients
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Shengdi Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1316-307
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — Pemetrexed; Carboplatin; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental)
  Interventions: Drug: Adebrelimab + SHR-8068 + Pemetrexed + Carboplatin
- Treatment group B (Active Comparator)
  Interventions: Drug: Camrelizumab + Pemetrexed + Carboplatin
- Treatment group C (Active Comparator)
  Interventions: Drug: Adebrelimab + Pemetrexed + Carboplatin

INTERVENTIONS:
Drug: Adebrelimab + SHR-8068 + Pemetrexed + Carboplatin — Adebrelimab,1200mg; SHR-8068, 1.0 mg/kg; Pemetrexed, 500mg/m2; Carboplatin, AUC 5 mg/mL/min
  Arms: Treatment group A
Drug: Camrelizumab + Pemetrexed + Carboplatin — Camrelizumab,200mg;Pemetrexed, 500mg/m2; Carboplatin, AUC 5 mg/mL/min
  Arms: Treatment group B
Drug: Adebrelimab + Pemetrexed + Carboplatin — Adebrelimab,1200mg; Pemetrexed, 500mg/m2; Carboplatin, AUC 5 mg/mL/min
  Arms: Treatment group C

SUMMARY:
Evaluating the Efficacy and safety of Adebrelimab in Combination with Platinum-based Doublet Chemotherapy and SHR-8068 as First-line Therapy for Patients with Advanced or Metastatic NSCLC Carrying STK11/KEAP1/KRAS Mutations

ELIGIBILITY:
Inclusion Criteria:

1. The participant voluntarily joins this clinical research study, understands the research procedures, and is capable of providing written informed consent by signing the Informed Consent Form.
2. At the time of signing the Informed Consent Form, participants must be between the ages of 18 and 75 years old (inclusive), with no gender restrictions.
3. Diagnosed with advanced or metastatic non-squamous NSCLC (non-small cell lung cancer) confirmed by histology or cytology.
4. At least one measurable tumor lesion outside the central nervous system that meets the RECIST v1.1guidelines .
5. The participant is expected to have a life expectancy of at least 12 weeks.
6. Participants must have tumors with STK11 or KEAP1 or KRAS mutations. Co-mutations are also allowed.
7. The participant must have adequate bone marrow and organ function.

Exclusion Criteria:

1. Pathologically or cytologically confirmed mixed Small Cell Lung Cancer (SCLC), sarcomatoid carcinoma, or neuroendocrine carcinoma.
2. Subjects with untreated or active Central Nervous System (CNS) metastases, those with a history of leptomeningeal metastasis, or those currently presenting with leptomeningeal metastasis.
3. Subjects with spinal cord compression that has not been radically treated by surgery and/or radiotherapy.
4. Subjects with inadequately controlled pain related to their tumor(s).
5. Subjects with a history of or concurrent other malignancies, except for basal cell carcinoma of the skin, superficial bladder cancer, cutaneous squamous cell carcinoma, in situ cervical cancer, localized prostate cancer, ductal carcinoma in situ following mastectomy (allowing for hormonal treatment for non-metastatic prostate or breast cancer), and papillary thyroid cancer which have achieved complete remission for at least 5 years prior to screening and do not require or are not expected to require further treatment during the study period.
6. Subjects who have received Chinese herbal anti-tumor treatment within 2 weeks prior to initiating the study treatment.
7. Subjects whose toxicities and/or complications from previous interventions have not resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE 5.0) Grade ≤1.
8. Subjects participating in another clinical study or whose initiation of study treatment is less than 4 weeks since the end of the last clinical study (last dose administration), or less than five half-lives of that study drug, whichever is shorter.
9. Subjects who have received systemic immunostimulant treatment within 4 weeks prior to starting the study treatment.
10. Subjects who have received systemic immunosuppressive treatment within 2 weeks prior to starting the study treatment.
11. Subjects with any active, known, or suspected autoimmune disease.
12. Subjects with severe heart disease.
13. Subjects who have experienced arterial or venous thrombotic events within 3 months prior to starting the study treatment.
14. Subjects with active syphilis infection.
15. Subjects who have had a severe infection within 4 weeks prior to starting the study treatment.
16. Subjects who have previously undergone or are planning to undergo allogeneic hematopoietic stem cell transplantation or organ transplantation.
17. Subjects with a history of severe hypersensitivity reactions to other monoclonal antibodies.
18. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study period.
19. Subjects with a history of substance abuse of psychoactive drugs, alcoholism, or drug addiction.
20. Subjects whom the investigator believes have any medical condition (such as pulmonary, metabolic, endocrine, or neurological diseases, congenital disorders, etc.), psychiatric conditions, or social circumstances that could potentially interfere with the subject's rights, safety, health, or ability to provide informed consent, cooperate, and participate in the study, or interfere with the assessment of the investigational drug, interpretation of subject safety data, or study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed Objective Response Rate (Phase One) | about 3 years
Overall Survival (Phase Two) | about 3.5 years

SECONDARY OUTCOMES:
The incidence and severity of Adverse Events (AEs) (Phases One and Two) | about 4.5 years
Duration of Response (DoR) based on Investigator Assessment (Phases One and Two) | about 6.5 years
Disease Control Rate (DCR) based on Investigator Assessment (Phases One and Two) | about 6.5 years
Progression-Free Survival (PFS) based on Investigator Assessment (Phases One and Two) | about 6.5 years
Overall Survival (OS) (Phase One) | about 3.5 years
Objective Response Rate (ORR) based on Investigator Assessment (Phase Two) | about 4.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Tumor Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided